CLINICAL TRIAL: NCT04008030
Title: A Phase 3 Randomized Clinical Trial of Nivolumab Alone, Nivolumab in Combination With Ipilimumab, or Investigator's Choice Chemotherapy in Participants With Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) Metastatic Colorectal Cancer
Brief Title: A Study of Nivolumab, Nivolumab Plus Ipilimumab, or Investigator's Choice Chemotherapy for the Treatment of Participants With Deficient Mismatch Repair (dMMR)/Microsatellite Instability High (MSI-H) Metastatic Colorectal Cancer (mCRC)
Acronym: CheckMate 8HW
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-8HW; 2018-000040-26 (EudraCT Number)
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Ipilimumab; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Bevacizumab; Cetuximab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Nivolumab Monotherapy (Experimental)
  Interventions: Biological: Nivolumab
- Arm B: Nivolumab + Ipilimumab Combination (Experimental)
  Interventions: Biological: Ipilimumab; Biological: Nivolumab
- Arm C: Investigator's Choice Chemotherapy (Active Comparator): Participants in Arm C would be allowed to receive Nivolumab + Ipilimumab if they progress
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Irinotecan; Drug: Bevacizumab; Drug: Cetuximab

INTERVENTIONS:
Biological: Ipilimumab — Specified dose on specified days
  Arms: Arm B: Nivolumab + Ipilimumab Combination
Drug: Oxaliplatin — Specified dose on specified days
  Arms: Arm C: Investigator's Choice Chemotherapy
Drug: Leucovorin — Specified dose on specified days
  Arms: Arm C: Investigator's Choice Chemotherapy
Drug: Fluorouracil — Specified dose on specified days
  Arms: Arm C: Investigator's Choice Chemotherapy
Drug: Irinotecan — Specified dose on specified days
  Arms: Arm C: Investigator's Choice Chemotherapy
Drug: Bevacizumab — Specified dose on specified days
  Arms: Arm C: Investigator's Choice Chemotherapy
Drug: Cetuximab — Specified dose on specified days
  Arms: Arm C: Investigator's Choice Chemotherapy
Biological: Nivolumab — Specified dose on specified days
  Arms: Arm A: Nivolumab Monotherapy; Arm B: Nivolumab + Ipilimumab Combination

SUMMARY:
The main purpose of this study is to compare the clinical benefit, as measured by Progression-Free Survival (PFS), Objective Response Rate (ORR), and Overall Survival (OS), achieved by nivolumab in combination with ipilimumab or by nivolumab monotherapy in participants with Microsatellite Instability High (MSI-H) or Mismatch Repair Deficient (dMMR) metastatic colorectal cancer (mCRC). This study will also compare nivolumab plus ipilimumab combination vs chemotherapy for treatment of MSI-H/dMMR mCRC participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic colorectal cancer (CRC) irrespective of prior treatment history with chemotherapy and/or targeted agents not amenable to surgery (Applicable only during Part 1 enrollment of the study)
* Histologically confirmed recurrent or metastatic CRC with no prior treatment history with chemotherapy and/or targeted agents for metastatic disease and not amenable to surgery (Applicable during Part 2 enrollment of the study)
* Known tumor microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) status per local standard of practice
* Eastern cooperative oncology group (ECOG) performance status lower than or equal to 1

Exclusion Criteria:

* An active, known or suspected autoimmune disease
* History of interstitial lung disease or pneumonitis
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2026-06-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (157):
- United States (9):
  - Local Institution - 0059, Los Angeles, California
  - Local Institution - 0130, Sacramento, California
  - Local Institution - 0103, Denver, Colorado
  - Local Institution - 0119, Arlington Heights, Illinois
  - Local Institution - 0060, New York, New York
  - Local Institution - 0105, Portland, Oregon
  - Local Institution - 0121, Pittsburgh, Pennsylvania
  - Local Institution - 0106, Dallas, Texas
  - Local Institution - 0104, Roanoke, Virginia
- Argentina (5):
  - Local Institution - 0073, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Local Institution - 0074, Viedma, Río Negro Province
  - Local Institution - 0084, Buenos Aires
  - Local Institution - 0100, CABA
  - Local Institution - 0072, CABA
- Australia (5):
  - Local Institution - 0019, Westmead, New South Wales
  - Local Institution - 0053, Woolloongabba, Queensland
  - Local Institution - 0018, Elizabeth Vale, South Australia
  - Local Institution - 0041, Clayton, Victoria
  - Local Institution - 0017, Heidelberg, Victoria
- Austria (5):
  - Local Institution - 0064, Graz
  - Local Institution - 0068, Linz
  - Local Institution - 0120, Salzburg
  - Local Institution - 0065, Vienna
  - Local Institution - 0067, Wiener Neustadt
- Belgium (3):
  - Local Institution - 0045, Bonheiden, Antwerpen
  - Local Institution - 0025, Anderlecht, Bruxelles-Capitale, Région de
  - Local Institution - 0024, Leuven
- Brazil (8):
  - Local Institution - 0096, Ipatinga, Minas Gerais
  - Local Institution - 0200, Natal, Rio Grande do Norte
  - Local Institution - 0192, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0102, Barretos, São Paulo
  - Local Institution - 0094, São José do Rio Preto, São Paulo
  - Local Institution - 0095, São Paulo, São Paulo
  - Local Institution - 0199, Rio de Janeiro
  - Local Institution - 0193, São Paulo
- Canada (5):
  - Local Institution - 0011, Edmonton, Alberta
  - Local Institution - 0039, Vancouver, British Columbia
  - Local Institution - 0013, Toronto, Ontario
  - Local Institution - 0016, Montreal, Quebec
  - Local Institution - 0015, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0070, Independencia, Santiago Metropolitan
  - Local Institution - 0071, Santiago, Santiago Metropolitan
  - Local Institution - 0069, Santiago, Santiago Metropolitan
- China (28):
  - Local Institution - 0146, Hefei, Anhui
  - Local Institution - 0163, Xiamen, Fujian
  - Local Institution - 0207, Zhangzhou, Fujian
  - Local Institution - 0211, Lanzhou, Gansu
  - Local Institution - 0158, Foshan, Guangdong
  - Local Institution - 0167, Guangzhou, Guangdong
  - Local Institution - 0153, Guangzhou, Guangdong
  - Local Institution - 0149, Guangzhou, Guangdong
  - Local Institution - 0160, Nanning, Guangxi
  - Local Institution - 0196, Nanning, Guangxi
  - Local Institution - 0180, Harbin, Heilongjiang
  - Local Institution - 0181, Zhengzhou, Henan
  - Local Institution - 0197, Changsha, Hunan
  - Local Institution - 0145, Changzhou, Jiangsu
  - Local Institution - 0151, Nanchang, Jiangxi
  - Local Institution - 0164, Changchun, Jilin
  - Local Institution - 0162, Shenyang, Liaoning
  - Local Institution - 0188, Xi'an, Shaanxi
  - Local Institution - 0210, Jinan, Shandong
  - Local Institution - 0212, Linyi, Shandong
  - Local Institution - 0154, Qingdao, Shandong
  - Local Institution - 0165, Yantai, Shandong
  - Local Institution - 0143, Shanghai, Shanghai Municipality
  - Local Institution - 0131, Shanghai, Shanghai Municipality
  - Local Institution - 0221, Shanghai, Shanghai Municipality
  - Local Institution - 0195, Kunming, Yunnan
  - Local Institution - 0137, Hangzhou, Zhejiang
  - Local Institution - 0206, Ningbo, Zhejiang
- Czechia (4):
  - Local Institution - 0087, Brno
  - Local Institution - 0085, Hradec Králové
  - Local Institution - 0088, Nový Jičín
  - Local Institution - 0086, Olomouc
- Denmark (2):
  - Local Institution - 0038, Herlev
  - Local Institution - 0036, Vejle
- France (14):
  - Local Institution - 0176, Limoges, Haute-Vienne
  - Local Institution - 0138, Lille, Nord
  - Local Institution - 0186, Bayonne
  - Local Institution - 0028, Besançon
  - Local Institution - 0183, Lyon
  - Local Institution - 0029, Lyon
  - Local Institution - 0066, Marseille
  - Local Institution - 0030, Montpellier
  - Local Institution - 0032, Nantes
  - Local Institution - 0027, Paris
  - Local Institution - 0061, Pessac
  - Local Institution - 0031, Poitiers
  - Local Institution - 0184, Strasbourg
  - Local Institution - 0040, Toulouse
- Germany (8):
  - Local Institution - 0042, Dresden
  - Local Institution - 0007, Essen
  - Local Institution - 0043, Hamburg
  - Local Institution - 0117, Hamburg
  - Local Institution - 0008, Hanover
  - Local Institution - 0009, Heidelberg
  - Local Institution - 0044, Marburg
  - Local Institution - 0010, Munich
- Greece (5):
  - Local Institution - 0222, Athens
  - Local Institution - 0123, Athens
  - Local Institution - 0124, Cholargós
  - Local Institution - 0125, Heraklion
  - Local Institution - 0126, Ioannina
- Ireland (3):
  - Local Institution - 0091, Dublin, Dublin
  - Local Institution - 0022, Dublin
  - Local Institution - 0026, Limerick
- Italy (6):
  - Local Institution - 0055, Catania
  - Local Institution - 0003, Genova
  - Local Institution - 0001, Milan
  - Local Institution - 0004, Napoli
  - Local Institution - 0002, Padua
  - Local Institution - 0054, Roma
- Japan (20):
  - Local Institution - 0109, Nagoya, Aichi-ken
  - Local Institution - 0112, Chiba, Chiba
  - Local Institution - 0107, Kashiwa-shi, Chiba
  - Local Institution - 0132, Matsuyama, Ehime
  - Local Institution - 0116, Fukuoka, Fukuoka
  - Local Institution - 0174, Sapporo, Hokkaido
  - Local Institution - 0128, Kanazawa, Ishikawa-ken
  - Local Institution - 0111, Kawasaki, Kanagawa
  - Local Institution - 0175, Yokohama, Kanagawa
  - Local Institution - 0133, Kumamoto, Kumamoto
  - Local Institution - 0189, Ōsaki, Miyagi
  - Local Institution - 0177, Kurashiki, Okayama-ken
  - Local Institution - 0115, Suita-shi, Osaka
  - Local Institution - 0187, Hidaka, Saitama
  - Local Institution - 0110, Kitaadachigun, Saitama
  - Local Institution - 0108, Sunto-gun, Shizuoka
  - Local Institution - 0118, Chuo-ku, Tokyo
  - Local Institution - 0113, Koto-ku, Tokyo
  - Local Institution - 0129, Minato-ku, Tokyo
  - Local Institution - 0114, Osaka
- Netherlands (3):
  - Local Institution - 0052, Amsterdam, North Holland
  - Local Institution - 0051, Amsterdam, North Holland
  - Local Institution - 0050, Utrecht
- Norway (3):
  - Local Institution - 0033, Bergen
  - Local Institution - 0034, Lorenskog
  - Local Institution - 0035, Oslo
- Local Institution - 0058, Rio Piedras, Puerto Rico
- Romania (6):
  - Local Institution - 0076, Cluj-Napoca, Cluj
  - Local Institution - 0081, Craiova, Dolj
  - Local Institution - 0168, Brasov
  - Local Institution - 0080, Bucharest
  - Local Institution - 0205, Iași
  - Local Institution - 0089, Suceava
- Spain (7):
  - Local Institution - 0056, Badalona, Barcelona [Barcelona]
  - Local Institution - 0173, A Coruña
  - Local Institution - 0006, Barcelona
  - Local Institution - 0005, Madrid
  - Local Institution - 0172, Málaga
  - Local Institution - 0063, Seville
  - Local Institution - 0171, Valencia
- Turkey (Türkiye) (2):
  - Local Institution - 0092, Adana
  - Local Institution - 0101, Istanbul
- United Kingdom (2):
  - Local Institution - 0127, London
  - Local Institution - 0049, Oxford

REFERENCES:
- [Derived] Andre T, Elez E, Lenz HJ, Jensen LH, Touchefeu Y, Van Cutsem E, Garcia-Carbonero R, Tougeron D, Mendez GA, Schenker M, de la Fouchardiere C, Limon ML, Yoshino T, Li J, Manzano Mozo JL, Dahan L, Tortora G, Chalabi M, Goekkurt E, Braghiroli MI, Joshi R, Cil T, Aubin F, Cela E, Chen T, Lei M, Jin L, Blum SI, Lonardi S. Nivolumab plus ipilimumab versus nivolumab in microsatellite instability-high metastatic colorectal cancer (CheckMate 8HW): a randomised, open-label, phase 3 trial. Lancet. 2025 Feb 1;405(10476):383-395. doi: 10.1016/S0140-6736(24)02848-4. Epub 2025 Jan 25. PMID 39874977
- [Derived] Andre T, Elez E, Van Cutsem E, Jensen LH, Bennouna J, Mendez G, Schenker M, de la Fouchardiere C, Limon ML, Yoshino T, Li J, Lenz HJ, Manzano Mozo JL, Tortora G, Garcia-Carbonero R, Dahan L, Chalabi M, Joshi R, Goekkurt E, Braghiroli MI, Cil T, Cela E, Chen T, Lei M, Dixon M, Abdullaev S, Lonardi S; CheckMate 8HW Investigators. Nivolumab plus Ipilimumab in Microsatellite-Instability-High Metastatic Colorectal Cancer. N Engl J Med. 2024 Nov 28;391(21):2014-2026. doi: 10.1056/NEJMoa2402141. PMID 39602630
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04008030.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Nivolumab Monotherapy: Nivolumab 240 mg infusion on Day 1 and every two weeks during cycles 1 and 2 for a total of 6 doses. Starting from Cycle 3 Day 1 participants received Nivolumab 480 mg infusion every 4 weeks.
- Arm B - Nivolumab + Ipilimumab: Nivolumab 240 mg infusion followed by Ipilimumab 1 mg/kg IV on Day 1 and every three weeks during cycles 1 and 2 for a total of 4 doses. Starting from Cycle 3 Day 1, participants received Nivolumab 480 mg infusion every 4 weeks.
- Arm C - Investigator's Choice Chemotherapy: Participants received standard of care chemotherapy
Period: Pre-Treatment
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Started (Randomized) | 353 | 354 | 132
Completed (Treated) | 351 | 352 | 115
Not Completed | 2 | 2 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 9
Not completed — Participant no longer meets study criteria | 2 | 1 | 2
Not completed — Other reasons | 0 | 1 | 6
Period: Treatment
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Started (Treated) | 351 | 352 | 115
Crossover to Arm B | 0 | 0 | 60
Completed | 137 | 159 | 0
Not Completed | 214 | 193 | 115
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Death | 2 | 4 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Participant no longer meets study criteria | 0 | 1 | 0
Not completed — Other reasons | 5 | 13 | 6
Not completed — Disease Progression | 137 | 82 | 85
Not completed — Study drug toxicity | 28 | 48 | 8
Not completed — Adverse Event unrelated to study drug | 28 | 22 | 6
Not completed — Maximum Clinical Benefit | 0 | 1 | 9
Not completed — On-going treatment | 13 | 20 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy | Total
Number analyzed (Participants) | 353 | 354 | 132 | 839
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (13.76) | 60.5 (13.14) | 61.3 (14.93) | 60.5 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 192 | 68 | 423
  Male | 190 | 162 | 64 | 416
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 32 | 11 | 77
  Not Hispanic or Latino | 189 | 165 | 67 | 421
  Unknown or Not Reported | 130 | 157 | 54 | 341
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 36 | 27 | 15 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 2 | 13
  White | 305 | 311 | 113 | 729
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 12 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) - Arm B vs. Arm A All Lines Centrally Confirmed MSI-H/dMMR
Description: BICR-assessed Progression-free survival (PFS) is defined as the time from the randomization date to the date of first objectively documented disease progression per RECIST 1.1 (i.e, radiologic) or death due to any cause, whichever occurs first.
Time Frame: From date of randomization to the date of first objectively documented disease progression or death due to any cause, whichever occurs first (Up to approximately 60 months)
Population: All randomized participants with centrally confirmed DNA mismatch repairdeficient/microsatellite instability-high metastatic colorectal cancer (dMMR/MSI-H mCRC) in Arm A and Arm B only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 286 | 296
Months | 39.26 [2.11 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | NA [53.82 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; p = 0.0003, Log Rank — Boundary for statistical significance p-value < 0.0095; Log-rank test stratified by the same factors as used in the Cox proportional hazard model; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.48 to 0.81] — a Cox Model stratified by tumor sidedness (left vs. right) and prior lines of therapy (0, 1, >= 2) as entered into the IRT

2. Primary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) - Arm B vs. Arm C 1L Participants Centrally Confirmed MSI-H/dMMR
Description: as for outcome 1
Time Frame: From date of randomization to the date of first objectively documented disease progression or death due to any cause, whichever occurs first (Up to approximately 32 months)
Population: All randomized participants with centrally confirmed DNA mismatch repairdeficient/microsatellite instability-high metastatic colorectal cancer (dMMR/MSI-H mCRC) who have not received prior therapy for metastatic disease (1L) in Arm B and Arm C only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Number analyzed (Participants) | 171 | 84
Months | NA [38.44 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | 5.85 [4.37 to 7.79]
Statistical Analysis 1: Comparison: Arm B - Nivolumab + Ipilimumab vs Arm C - Investigator's Choice Chemotherapy; Test type: Superiority — Arm B over Arm C; p < 0.0001, Log Rank — Boundary for statistical significance p-value < 0.0209; Log-rank test stratified by the same factors as used in the Cox proportional hazard model; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.14 to 0.32] — From a Cox Model stratified by tumor sidedness (left vs. right) as entered into the IRT

3. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) - 1L Participants
Description: as for outcome 1
Time Frame: From date of randomization to the date of first objectively documented disease progression or death due to any cause, whichever occurs first
Reporting Status: Not Posted, anticipated posting 2027-05

4. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) - Arm B vs. Arm A All Randomized Participants
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants in Arm A and Arm B only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 353 | 354
Months | 18.43 [9.20 to 28.16] | 54.08 [44.02 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.52 to 0.79] — from a Cox Model stratified by tumor sidedness (left vs. right) and prior lines of therapy (0, 1, >= 2) as entered into the IRT

5. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) - 1L Randomized Participants
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants who have not received prior therapy for metastatic disease (1L)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Number analyzed (Participants) | 201 | 202 | 101
Months | 44.85 [18.23 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | NA [34.30 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | 6.21 [4.70 to 9.00]
Statistical Analysis 1: Comparison: Arm B - Nivolumab + Ipilimumab vs Arm C - Investigator's Choice Chemotherapy; Test type: Superiority — Arm B over Arm C; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.23 to 0.46] — From a Cox Model stratified by tumor sidedness (left vs. right) as entered into the IRT

6. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) - Crossover and First Line Arm
Description: as for outcome 1
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2027-05

7. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) by Polymerase Chain Reaction (PCR) - Arm B vs. Arm A
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants with centrally confirmed microsatellite instability-high (MSI-H) in Arm A and Arm B only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 246 | 257
Months | NA [24.80 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | NA [53.82 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Hazard Ratio (HR) = 0.60, 95% CI [0.45 to 0.80] — from a Cox proportional hazard model stratified by tumor sidedness (left vs right) and prior lines of therapy (0, 1, ≥ 2) per IRT

8. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) by Immunohistochemistry (IHC) - Arm B vs. Arm A
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants with centrally confirmed DNA mismatch repairdeficient (dMMR) in Arm A and Arm B only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 271 | 280
Months | 44.29 [25.56 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | NA [53.82 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Hazard Ratio (HR) = 0.63, 95% CI [0.48 to 0.83] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) by Polymerase Chain Reaction (PCR) - Arm B vs. Arm C
Description: as for outcome 1
Time Frame: as for outcome 2
Population: All randomized participants with centrally confirmed microsatellite instability-high (MSI-H) who have not received prior therapy for metastatic disease (1L) in Arm B and Arm C only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Number analyzed (Participants) | 147 | 71
Months | NA [38.44 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | 6.21 [4.70 to 9.03]
Statistical Analysis 1: Comparison: Arm B - Nivolumab + Ipilimumab vs Arm C - Investigator's Choice Chemotherapy; Test type: Superiority — Arm B over Arm C; Hazard Ratio (HR) = 0.20, 95% CI [0.12 to 0.31] — From a stratified Cox proportional hazard model by tumor sidedness (left vs. right) as entered into the IRT

10. Secondary Outcome: Progression-free Survival (PFS) by Blinded Independent Review Center (BICR) by Immunohistochemistry (IHC) - Arm B vs. Arm C
Description: as for outcome 1
Time Frame: as for outcome 2
Population: All randomized participants with centrally confirmed DNA mismatch repairdeficient (dMMR) who have not received prior therapy for metastatic disease (1L) in Arm B and Arm C only
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Number analyzed (Participants) | 147 | 71
Months | NA [38.44 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | 6.21 [4.70 to 9.03]
Statistical Analysis 1: Comparison: Arm B - Nivolumab + Ipilimumab vs Arm C - Investigator's Choice Chemotherapy; Test type: Superiority — Arm B over Arm C; Hazard Ratio (HR) = 0.20, 95% CI [0.12 to 0.31] — From a stratified Cox proportional hazard model by tumor sidedness (left vs. right) as entered into the IRT

11. Secondary Outcome: Progression-free Survival (PFS) by Investigator- Arm B vs. Arm A All Lines
Description: Investigator-assessed Progression-free survival (PFS) is defined as the time from the randomization date to the date of first objectively documented disease progression per RECIST 1.1 (i.e, radiologic) or death due to any cause, whichever occurs first.
Time Frame: as for outcome 1
Population: All randomized participants in Arm A and Arm B only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 353 | 354
Months | 22.18 [11.70 to 29.44] | 54.08 [41.17 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Hazard Ratio (HR) = 0.64, 95% CI [0.52 to 0.79] — [estimate comment as in outcome 4, analysis 1]

12. Secondary Outcome: Progression-free Survival (PFS) by Investigator - Arm A and Arm B All Lines With dMMR/MSI-H mCRC
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 286 | 296
Months | 38.14 [27.20 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | NA [54.08 to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Hazard Ratio (HR) = 0.62, 95% CI [0.48 to 0.80] — Cox Model stratified by tumor sidedness (left vs. right) and prior lines of therapy (0, 1, >= 2) as entered into the IRT

13. Secondary Outcome: Progression-free Survival (PFS) by Investigator - 1L Participants
Description: as for outcome 11
Time Frame: From date of randomization to the date of first objectively documented disease progression or death due to any cause, whichever occurs first (Up to approximately 60 months for arm A and arm B; up to 32 months for arm C)
Reporting Status: Not Posted, anticipated posting 2027-05

14. Secondary Outcome: Objective Response Rate (ORR) by Blinded Independent Review Center (BICR) - Arm A and Arm B All Lines With dMMR/MSI-H mCRC
Description: Objective Response Rate (ORR) is defined as the percentage of all randomized participants whose best overall response is either confirmed complete response (CR) or confirmed partial response (PR).
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive disease (PD)=At least a 20% increase in the sum of diameters of target lesions. the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From date of randomization to the date of the initial objectively documented tumor progression, or the date of initiation of subsequent therapy, whichever occurs first (Up to approximately 60 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 286 | 296
Percentage of participants | 57.7 [51.7 to 63.5] | 70.6 [65.1 to 75.7]
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; p = 0.0011, Cochran-Mantel-Haenszel — Boundary for statistical significance p-value < 0.006; Two-sided p-value from stratified CMH Test; Odds Ratio (OR) = 1.77, 95% CI [1.26 to 2.50]; Stratified by tumor sidedness (left vs. right) and prior lines of therapy (0, 1, >= 2) as entered into the IRT

15. Secondary Outcome: Objective Response Rate (ORR) by Blinded Independent Review Center (BICR) - 1L Participants
Description: as for outcome 14
Time Frame: as for outcome 14
Population: All randomized participants with centrally confirmed DNA mismatch repairdeficient/microsatellite instability-high metastatic colorectal cancer (dMMR/MSI-H mCRC) who have not received prior therapy for metastatic disease (1L)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab | Arm C - Investigator's Choice Chemotherapy
Number analyzed (Participants) | 170 | 171 | 84
Percentage of participants | 61.2 [53.4 to 68.5] | 72.5 [65.2 to 79.1] | 27.4 [18.2 to 38.2]
Statistical Analysis 1: Comparison: Arm B - Nivolumab + Ipilimumab vs Arm C - Investigator's Choice Chemotherapy; Test type: Superiority — Arm B over Arm C; Odds Ratio (OR) = 7.02, 95% CI [3.91 to 12.62] — Stratified by tumor sidedness (left vs. right)
Statistical Analysis 2: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Odds Ratio (OR) = 1.67, 95% CI [1.06 to 2.63] — Stratified by tumor sidedness (left vs. right)

16. Secondary Outcome: Overall Survival (OS) - Arm B vs. Arm A All Lines With dMMR/MSI-H mCRC
Description: Overall Survival (OS) is defined as the time from the randomization date to the date of death due to any cause. A participant who has not died will be censored at last known date alive.
Time Frame: From randomization to the date of death due to any cause (Up to approximately 60 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Nivolumab Monotherapy | Arm B - Nivolumab + Ipilimumab
Number analyzed (Participants) | 286 | 296
Months | NA [NA to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates | NA [NA to NA] — Insufficient number of participants with events based on Kaplan-Meier Estimates
Statistical Analysis 1: Comparison: Arm A - Nivolumab Monotherapy vs Arm B - Nivolumab + Ipilimumab; Test type: Superiority — Arm B over Arm A; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.45 to 0.83] — [estimate comment as in outcome 4, analysis 1]

17. Secondary Outcome: Overall Survival (OS) - 1L Participants
Description: as for outcome 16
Time Frame: From randomization to the date of death due to any cause
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their primary completion (up to approximately 60 months). SAEs and Other AEs were assessed from first dose up to 100 days post last dose (Up to approximately 60 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Arm A: Nivolumab: Nivolumab 240 mg infusion on Day 1 and every two weeks during cycles 1 and 2 for a total of 6 doses. Starting from Cycle 3 Day 1 participants received Nivolumab 480 mg infusion every 4 weeks.
- Arm B: Nivolumab + Ipilimumab: Nivolumab 240 mg infusion followed by Ipilimumab 1 mg/kg IV on Day 1 and every three weeks during cycles 1 and 2 for a total of 4 doses. Starting from Cycle 3 Day 1, participants received Nivolumab 480 mg infusion every 4 weeks.
- Arm C: Chemotherapy: Participants received standard of care chemotherapy
- Crossover: Nivolumab + Ipilimumab: Participants assigned to Arm C that experience documented progression of disease (PD) per RECIST 1.1 by Blinded Independent Central Review (BICR) will have an option to crossover to nivolumab plus ipilimumab therapy (Arm B)
Arm/Group | Arm A: Nivolumab | Arm B: Nivolumab + Ipilimumab | Arm C: Chemotherapy | Crossover: Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 150/353 | 103/354 | 62/132 | 24/60
Serious Adverse Events (participants affected / at risk) | 161/351 | 174/352 | 58/115 | 38/60
Other Adverse Events (participants affected / at risk) | 311/351 | 330/352 | 114/115 | 52/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab (N=351) | Arm B: Nivolumab + Ipilimumab (N=352) | Arm C: Chemotherapy (N=115) | Crossover: Nivolumab + Ipilimumab (N=60)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 2 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0 | 0
Sinoatrial block (Cardiac disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 4 | 11 | 0 | 2
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 3 | 10 | 0 | 2
Hypopituitarism (Endocrine disorders) | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0
Primary adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 7 | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 5 | 1 | 2
Colonic fistula (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 8 | 4 | 3
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhagic necrotic pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 7 | 0 | 4 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 2 | 6 | 0 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 9 | 6 | 6 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 4 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 7 | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 5 | 1 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1 | 2
Asthenia (General disorders) | 2 | 2 | 2 | 0
Complication of device insertion (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Device related thrombosis (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
General physical health deterioration (General disorders) | 6 | 1 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Inadequate analgesia (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Multi-organ disorder (General disorders) | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Obstruction (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 3 | 2 | 1
Sudden death (General disorders) | 0 | 2 | 0 | 1
Ulcer (General disorders) | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 3 | 2 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0 | 2
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 2 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Abdominal infection (Infections and infestations) | 2 | 1 | 1 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 6 | 3 | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium colitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 2 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
HIV infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 2 | 2 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 2
Klebsiella urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 1 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 7 | 4 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 6 | 4 | 0 | 2
Septic shock (Infections and infestations) | 3 | 4 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 4 | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 2 | 1 | 0 | 0
Vascular access site infection (Infections and infestations) | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 2 | 3 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urostomy complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 0
Clostridium test positive (Investigations) | 0 | 1 | 0 | 0
Cortisol decreased (Investigations) | 0 | 0 | 0 | 1
General physical condition abnormal (Investigations) | 2 | 5 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Postprandial hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 2 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 | 22 | 8 | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Acute polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Device breakage (Product Issues) | 1 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 2 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 6 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 0 | 0
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 2 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Loss of personal independence in daily activities (Social circumstances) | 0 | 1 | 0 | 0
Cancer surgery (Surgical and medical procedures) | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0 | 1
Embolism (Vascular disorders) | 1 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Jugular vein embolism (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0
Venous occlusion (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivolumab (N=351) | Arm B: Nivolumab + Ipilimumab (N=352) | Arm C: Chemotherapy (N=115) | Crossover: Nivolumab + Ipilimumab (N=60)
Anaemia (Blood and lymphatic system disorders) | 71 | 58 | 26 | 11
Neutropenia (Blood and lymphatic system disorders) | 3 | 10 | 26 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5 | 11 | 0
Adrenal insufficiency (Endocrine disorders) | 9 | 30 | 0 | 3
Hyperthyroidism (Endocrine disorders) | 18 | 43 | 1 | 4
Hypothyroidism (Endocrine disorders) | 35 | 65 | 1 | 9
Abdominal pain (Gastrointestinal disorders) | 67 | 64 | 31 | 9
Abdominal pain upper (Gastrointestinal disorders) | 20 | 27 | 7 | 6
Constipation (Gastrointestinal disorders) | 39 | 57 | 24 | 4
Diarrhoea (Gastrointestinal disorders) | 102 | 119 | 66 | 18
Dry mouth (Gastrointestinal disorders) | 18 | 22 | 2 | 3
Nausea (Gastrointestinal disorders) | 58 | 72 | 55 | 15
Stomatitis (Gastrointestinal disorders) | 14 | 9 | 12 | 1
Vomiting (Gastrointestinal disorders) | 38 | 39 | 27 | 7
Asthenia (General disorders) | 84 | 93 | 45 | 12
Fatigue (General disorders) | 67 | 70 | 23 | 11
Mucosal inflammation (General disorders) | 6 | 9 | 7 | 1
Oedema peripheral (General disorders) | 31 | 38 | 11 | 4
Pyrexia (General disorders) | 48 | 43 | 12 | 5
COVID-19 (Infections and infestations) | 32 | 42 | 6 | 8
Nasopharyngitis (Infections and infestations) | 11 | 19 | 4 | 1
Urinary tract infection (Infections and infestations) | 23 | 30 | 11 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 11 | 6 | 1
Alanine aminotransferase increased (Investigations) | 33 | 43 | 7 | 3
Amylase increased (Investigations) | 19 | 21 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 33 | 39 | 5 | 2
Blood alkaline phosphatase increased (Investigations) | 22 | 18 | 2 | 0
Blood bilirubin increased (Investigations) | 21 | 20 | 1 | 0
Blood creatinine increased (Investigations) | 17 | 22 | 3 | 5
Lipase increased (Investigations) | 18 | 26 | 4 | 6
Neutrophil count decreased (Investigations) | 6 | 5 | 19 | 2
Platelet count decreased (Investigations) | 10 | 3 | 8 | 0
Weight decreased (Investigations) | 19 | 20 | 12 | 4
White blood cell count decreased (Investigations) | 5 | 3 | 8 | 0
Decreased appetite (Metabolism and nutrition disorders) | 46 | 53 | 33 | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 11 | 6 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 22 | 19 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 12 | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 19 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 54 | 70 | 5 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 44 | 15 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 22 | 1 | 3
Dizziness (Nervous system disorders) | 12 | 17 | 4 | 4
Headache (Nervous system disorders) | 32 | 42 | 10 | 7
Neuropathy peripheral (Nervous system disorders) | 5 | 3 | 15 | 1
Neurotoxicity (Nervous system disorders) | 1 | 2 | 8 | 0
Paraesthesia (Nervous system disorders) | 4 | 6 | 10 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 7 | 8 | 2
Insomnia (Psychiatric disorders) | 17 | 25 | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 34 | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35 | 23 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 11 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 12 | 12 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 24 | 2 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 7 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 81 | 105 | 6 | 15
Rash (Skin and subcutaneous tissue disorders) | 40 | 45 | 9 | 6
Hypertension (Vascular disorders) | 24 | 26 | 14 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04008030/Prot_SAP_000.pdf